CLINICAL TRIAL: NCT01622816
Title: Prospective Determination of Agreement Between Standard ETDRS (Early Treatment Diabetic Retinopathy Study) Chart and Handheld Illuminated ETDRS Equivalent Chart in Eyes With Retinal Pathology
Brief Title: Comparing Visual Acuity Measurements (How Well You Can See) Using a Standard ETDRS Chart & a Handheld ETDRS Chart
Status: Completed | Type: Observational
Sponsor: Julia Haller (Other)
Responsible Party: Sponsor-Investigator, Julia Haller, Investigator, Wills Eye
Organization: Wills Eye (Other)
Other Study IDs: ETDRS2012
Record Dates: First submitted 2012-04-19; First posted 2012-06-19 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparing visual acuity measurements (measurements of how well you can see) using a standard ETDRS (Early Treatment Diabetic Retinopathy Study) chart and a handheld ETDRS chart

DETAILED DESCRIPTION:
Prospective determination of agreement between standard ETDRS chart and handheld illuminated ETDRS equivalent chart in eyes with retinal pathology

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and comply with study assessments for the full duration of the study (one visit per patient).
2. Age greater than 18 years.
3. Clinical diagnosis of retinal disease (including age-related macular degeneration, macular degeneration, retinal vessel occlusion, among others).

Exclusion Criteria:

1. Presence of a significant cataract as determined by your doctor.
2. Presence of a significant posterior capsular opacity (haziness in your eyes) as determined by your doctor.
3. Diagnosis of uveitis (inflammation in part of the eye).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in clinical trials for various retinal diseases at the Wills Eye Institute
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
ETDRS Letter Score | 1 Day
  To determine the visual acuity measurement using this handheld internally illuminated ETDRS chart, and a standard back illuminated EDTRS chart. This will be done during the visual acuity test.

SECONDARY OUTCOMES:
ETDRS Letter Score Consistency | 1 Day
  To use the score results to determine whether this new, handheld chart, called the RAM-ETDRS chart, is just as efficient as the standard ETDRS eye chart in measuring your vision. This will be done during your visual acuity exam.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Haller, MD, Principal Investigator — Wills Eye Institute
Locations (1):
- Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahimy E, Reddy S, DeCroos FC, Khan MA, Boyer DS, Gupta OP, Regillo CD, Haller JA. PROSPECTIVE EVALUATION OF VISUAL ACUITY AGREEMENT BETWEEN STANDARD EARLY TREATMENT DIABETIC RETINOPATHY STUDY CHART AND A HANDHELD EQUIVALENT IN EYES WITH RETINAL PATHOLOGY. Retina. 2015 Aug;35(8):1680-7. doi: 10.1097/IAE.0000000000000518. PMID 25719987